CLINICAL TRIAL: NCT07058883
Title: Prospective, Randomized, Placebo-Controlled, Multicenter Clinical Trial Evaluating the Efficacy and Safety of Juläine (Polylactic Acid) in the Treatment of Facial Acne Scars
Brief Title: Evaluation of Juläine (TM) for the Treatment of Atrophic Facial Acne Scars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordberg Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB 15-TF-EU-100-04F
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acne Scars
Keywords: polylactic acid; facial scars; acne; aesthetic; injectable device
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juläine Group (Experimental): Participants in this arm will receive three intradermal injections of Juläine, an injectable polylactic acid gel, at Day 0, Day 30, and Day 60. Injections are administered into areas affected by atrophic acne scars.
  Interventions: Device: Juläine
- Placebo Group (Placebo Comparator): Participants in this arm will receive three intradermal injections of sterile saline (placebo) at Day 0, Day 30, and Day 60, into areas affected by acne scars.
  Interventions: Other: Sterile Saline (Placebo)

INTERVENTIONS:
Device: Juläine — Juläine is a sterile injectable implant containing poly-L-lactic acid microspheres, intended for intradermal use to improve skin depressions from acne scars.
  Arms: Juläine Group
Other: Sterile Saline (Placebo) — Sterile saline solution used as a placebo control, administered in the same volume and schedule as Juläine.
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate the effectiveness and safety of Juläine, an injectable medical device made of polylactic acid, for treating facial acne scars. Participants with atrophic acne scars will be randomly assigned to receive either Juläine or a placebo (saline). The treatment will consist of three injection sessions over two months, followed by a 12-month observation period. The study will measure changes in scar severity and skin quality over time using clinical assessments and imaging tools. The study is being conducted at multiple dermatology clinics in Poland and is approved by a local ethics committee.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy and safety of Juläine, a sterile injectable medical device composed of polylactic acid microspheres in a carboxymethylcellulose gel, for the treatment of moderate to severe facial atrophic acne scars.

A total of 55 adult participants will be enrolled across selected dermatology sites in Poland. Forty-five participants will be randomized to receive Juläine, and ten participants will be randomized to receive a placebo (sterile saline solution). All participants will receive three treatment sessions administered over a two-month period (Day 0, Day 30, and Day 60), with injections targeted to areas affected by atrophic scars.

The primary endpoint is the improvement in acne scars at 12 months from baseline, assessed by blinded evaluators using the Acne Scar Rating Scale (ASRS). Secondary outcomes include subject-reported satisfaction, improvement assessments using the Global Aesthetic Improvement Scale (GAIS), and objective skin texture measurements evaluated through imaging systems such as Canfield VISIA.

Safety will be monitored through the collection of adverse events, local tolerability assessments, and follow-up visits over a 12-month period. The study is conducted in compliance with ISO 14155:2020 and EU MDR regulations, and has received ethics approval from the Bioethics Committee of the Regional Medical Chamber in Gdańsk, Poland.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presence of moderate to severe atrophic facial acne scars
* Immune-competent adult
* Willing and able to comply with study procedures and follow-up visits
* Signed informed consent obtained

Exclusion Criteria:

* Active acne, infection, or chronic skin disease in the treatment area
* Known allergy or hypersensitivity to any component of Juläine
* History of keloid formation or hypertrophic scarring
* Current anticoagulant therapy or bleeding disorder
* Pregnant or breastfeeding
* Previous aesthetic treatment in the same area within the past 6 months
* Participation in another interventional clinical trial within 30 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Average change in Acne Scar Rating Scale (ASRS) score from baseline to 6 and 12 months after treatment | 12 months after treatment
  Average change in ASRS score (scale 1-4; higher scores indicate worse scarring) from baseline to 6 and 12 months, assessed by blinded evaluators using photographs.

SECONDARY OUTCOMES:
Change in skin elasticity and hydration measured by cutometry | 3, 6, 9, and 12 months after treatment
  Elasticity is expressed in millimeters of skin retraction, with higher values indicating greater elasticity.
  Hydration is expressed in arbitrary units (AU), with higher values indicating greater hydration.
Global improvement based on GAIS evaluated by investigator and patient | 3, 6, 9, and 12 months after treatment
  GAIS is a 5-point ordinal scale:
  1. = Very much improved
  2. = Much improved
  3. = Improved
  4. = No change
  5. = Worse
  Lower scores indicate better aesthetic improvement.
Change in scar structure using high-frequency ultrasound (HFUS) | 12 months after treatment
  Scar depth is measured in millimeters (mm) via HFUS imaging with higher values indicating worse skin condition (more visible features).
Change in skin characteristics evaluated by VISIA imaging | Baseline, 6 months, and 12 months
  Skin features assessed using Canfield VISIA focusing on texture, pigmentation, and pores.
  Scores range from 0 to 100, with higher values indicating worse skin condition (more visible features).

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Individual Specialist Medical Practice Maria Luiza-Piesiaków, Gdansk
  - Centrum Medyczne dr Kubik, Gdynia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participant confidentiality and in compliance with data protection regulations. The study results will be disseminated in aggregate form through peer-reviewed publication and regulatory submissions, ensuring transparency while safeguarding privacy.